CLINICAL TRIAL: NCT00279890
Title: Proof of Concept Trial:SR-01 for the Treatment of Rosacea
Brief Title: Topical Agent for Treatment of Red Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Mark V. Dahl, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44-05; MCS 385
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Rosacea; Bilaterally Symmetric Red Skin on Cheeks
MeSH Terms: conditions — Rosacea

INTERVENTIONS:
Drug: Topical SR-01

SUMMARY:
SR-01 may reduce facial redness. it is a topically applied product. The agent will be applied to local skin areas of subjects with red facial skin to assess affect, and then applied to the whole face to assess efficacy and safety

ELIGIBILITY:
Bilaterally symmetric red skin on cheeks Caucasian Age 18-60 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Reduction of redness

SECONDARY OUTCOMES:
Safety and tolerability
Cosmetic acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Mark V. Dahl, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States